CLINICAL TRIAL: NCT00700648
Title: A Multicenter, Open Label, Nonrandomized, Non Interventional, Observational, Safety and Efficacy Study in Hospitalized Subjects Using Intravenous NovoRapid® (Insulin Aspart)
Brief Title: An Observational Study to Assess Safety and Effectiveness of Intravenous NovoRapid® in Hospitalised Subjects
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-3531
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Intravenous NovoRapid dose & frequency as decided by treating physician

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the side effects profile and benefits of using intravenous insulin aspart infusion in hospitalised subjects under normal clinical practice conditions in India.

ELIGIBILITY:
Inclusion Criteria:

* Any hospitalized subject with hyperglycaemia requiring intravenous insulin therapy is eligible for the study based on the discretion of the physician.

Exclusion Criteria:

* Subjects who are unlikely to comply with protocol, e.g., uncooperative attitude;
* Subjects with a hypersensitivity to NovoRapid or to any of the excipients.
* Subjects with conditions considered as contraindications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized subjects requiring intravenous insulin therapy
Sampling Method: Non-Probability Sample
Enrollment: 3024 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs (adverse event) | After 6 months
Incidence of SAEs (serious adverse event) | After 6 months

SECONDARY OUTCOMES:
Other safety & efficacy measures | After 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

REFERENCES:
- [Result] Intravenous insulin aspart in a hospital setting: results from an observational study examining patient outcomes and physician preferences; Udwadia F, Bhattacharyya A, Seshiah V et al.; Diabetes Manage. (2012) 2(2), 103-110
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com